CLINICAL TRIAL: NCT05030987
Title: Renal Denervation to Treat Heart Failure With Preserved Ejection Fraction - A Pilot Trial
Brief Title: Renal Denervation to Treat Heart Failure With Preserved Ejection Fraction
Acronym: UNLOAD-HFpEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: ReCor Medical, Inc. (Industry)
Responsible Party: Principal Investigator, Karl Fengler, PhD, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNLOAD-HFpEF; CIV-20-10-034846 (Other: Eudamed-Nr.)
Record Dates: First submitted 2021-08-30; First posted 2021-09-01 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Hypertension, Renal
Keywords: Renal Denervation; Hypertension; Heart Failure with Preserved Ejection Fraction
MeSH Terms: conditions — Hypertension, Renal; Hypertension | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RDN (Experimental): Renal Denervation
  Interventions: Procedure: Renal Denervation
- Sham (Sham Comparator): Sham Procedure
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: Renal Denervation — Renal denervation in patients with HFpEF and uncontrolled hypertension
  Arms: RDN
Procedure: Sham — Sham Treatment. After six months, cross-over is planned in all sham-treated patients and this patients will also receive a renal denervation.
  Other Names: Sham Procedure
  Arms: Sham

SUMMARY:
Heart failure with preserved ejection fraction has a high mortality, which is contrasted by a total absence of therapy options besides symptomatic diuretic treatment. This study aims to explore the potential of renal denervation as a treatment option for heart failure with preserved ejection fraction.

DETAILED DESCRIPTION:
Heart failure is one of the most important diseases worldwide, with a 5-year mortality of up to 75% in symptomatic patients. While substantial progress has been made in the treatment of patients with reduced left ventricular ejection fraction (HFrEF), mortality for patients with heart failure and preserved ejection fraction (HFpEF) remains unchanged, despite a comparable prevalence and mortality of the disease as for heart failure with reduced ejection fraction.

HFpEF is a heterogeneous condition and has been a diagnostic and therapeutic challenge for clinicians and researchers over the past decades. While some rare cases of HFpEF can be attributed to specific diseases like amyloidosis, in most other patients common characteristics are increased ventricular filling pressures and ventricular and arterial stiffening as frequently caused by ageing, diabetes and arterial hypertension. Furthermore, increased sympathetic activity has been described as one pathogenic contributor to chronic heart failure and is associated with poor clinical prognosis. It also leads to a more pulsatile BP profile which can cause a mismatch in arterio-ventricular coupling.

The modulating effects on the sympathetic nervous system induced by renal denervation (RDN) should be beneficial in HFpEF, as they improve resting and exercise hemodynamics due to an improved ventriculoarterial coupling by reduced aortic stiffness and lower systemic blood pressure. In addition, RDN leads to optimized stroke volume and stroke work and might affect cardiac preload by improving blood distribution into the splanchnic compartment.

This study aims to explore the potential of RDN as a therapy for HFpEF in a single center pilot trial using a randomized, sham-controlled double-blind design.

ELIGIBILITY:
Inclusion Criteria:

1. confirmed arterial hypertension (1-5 antihypertensive drugs without any dosage change in the preceding 4 weeks) and average systolic BP between >125 and ≤170 mmHg and diastolic BP ≤110 mmHg in 24h ambulatory blood pressure measurement (ABPM)
2. HFpEF (defined by clinical signs and/or symptoms of heart failure, objective structural cardiac abnormalities according to the ESC (European Society of Cardiology) criteria [1], elevated NT-proBNP ≥125 pg/mL and left-ventricular ejection fraction ≥55%)
3. NYHA-Class II or III
4. Confirmation of an elevated cardiac filling pressures (either LVEDP >= 16 mmHg or PCWP >= 15 mmHg at rest or >=25 mmHg during exercise) by catheterization
5. Age 18-80 years
6. Written informed consent

Exclusion Criteria:

1. ≥1 main renal artery diameter <3.0 mm
2. main renal artery length < 20 mm
3. a single functioning kidney
4. presence of abnormal kidney tumors
5. renal artery aneurysm
6. pre-existing renal stent or history of renal artery angioplasty
7. fibromuscular disease of the renal arteries
8. presence of renal artery stenosis of any origin ≥50%
9. iliac/femoral artery stenosis precluding femoral access for RDN
10. fertile women (within two years of their last menstruation) without appropriate contraceptive measures (implanon, injections, oral contraceptives, intrauterine devices, partner with vasectomy) while participating in the trial (participants using a hormone-based method have to be informed of possible effects of the trial device on contraception).
11. participation in other interventional trials
12. patients under legal supervision or guardianship
13. suspected lack of compliance
14. pregnant women
15. Presence of intracardiac pacemakers or implantable cardioverter/defibrillators

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
exercise pulmonary capillary wedge pressure (PCWP) at 20 W workload | 6 months after randomization
  To assess the hemodynamic effects of RDN in patients with HFpEF in comparison to sham-treatment

SECONDARY OUTCOMES:
number of combination of death, increase in diuretic therapy, hospitalization for heart failure, worsening NYHA-class, change in pulmonary pressure parameters | 6, 12 and 24 months after RDN
  number of combined endpoint in RDN and SHAM patients
Change in mean Pulmonary artery (PA) pressure, estimated pulmonary artery diastolic pressure (ePAD) and PA pressure variability from pulmonary pressure sensor measurements | 6 months after randomization
  difference between RDN and sham
Change in mean PA pressure, ePAD and PA pressure variability from pulmonary pressure sensor measurements | 6, 12 and 24 months after RDN
  Change in mean PA pressure, ePAD and PA pressure variability from pulmonary pressure sensor measurements, compared to baseline values
Change in Systolic/Diastolic 24h blood pressure by ABPM and blood pressure variability | 6 months after randomization
  difference between RDN and sham
Change in Systolic/Diastolic 24h blood pressure by ABPM and blood pressure variability | 6, 12 and 24 months after RDN
  Change in Systolic/Diastolic 24h blood pressure by ABPM and blood pressure variability, compared to baseline values
Difference in ventriculo-arterial coupling | 6 months after randomization
  Difference in ventriculo-arterial coupling (by end-systolic elastance and arterial elastance) as acquired by invasive measurement
Change in Cardiac magnetic resonance (CMR) based hemodynamics | 6 months after randomization
  Change in CMR-based hemodynamics (difference between RDN and sham) as compared to baseline values
Change in ventriculo-arterial coupling | 6 months after randomization
  Change in ventriculo-arterial coupling (cMRI and echocardiogram) (difference between RDN and sham) as compared to baseline values
Difference in resting and exercise PCWP (at 20, 40, 60, 80 W, and maximum workload) | 6 months after randomization
  Difference in resting and exercise PCWP (at 20, 40, 60, 80 W, and maximum workload) (difference between RDN and sham) as compared to baseline values
Difference in peak PCWP | 6 months after randomization
  Difference in peak PCWP (difference between RDN and sham) as compared to baseline values
Difference in NT-proBNP | 6 months after randomization
  Difference in NT-proBNP (difference between RDN and sham) as compared to baseline
Difference in NT-proBNP | 6, 12 and 24 months after RDN
  Difference in NT-proBNP as compared to baseline
number of patients with Hospitalizations for heart failure | 6 months after randomization
  number of patients with Hospitalizations for heart failure (difference between RDN and sham)
difference in All-cause Mortality | 6 months after randomization
  All-cause Mortality (difference between RDN and sham)
difference in cardiac mortality | 6 months after randomization
  cardiac mortality (difference between RDN and sham)
difference in major adverse cardiovascular events | 6 months after randomization
  major adverse cardiovascular events (composite of cardiac death, myocardial infarction, stroke and hospitalization for heart failure) (difference between RDN and sham)
difference in number of Adverse Events | 6 months after randomization
  Adverse events (difference between RDN and sham)
difference in Frequency of patients with controlled hypertension | 6 months after randomization
  Frequency of patients with controlled hypertension (blood pressure within treatment goals in ABPM as recommended by the European Society of Cardiology) (difference between RDN and sham)
difference in Frequency of patients with controlled hypertension | 6, 12 and 24 months after RDN
  Frequency of patients with controlled hypertension (blood pressure within treatment goals in ABPM as recommended by the European Society of Cardiology) as compared to baseline
Difference in 6-minute walk distance | 6 months after randomization
  Difference in 6-minute walk distance (difference between RDN and sham)
Difference in 6-minute walk distance | 6, 12 and 24 months after RDN
  Difference in 6-minute walk distance as compared to baseline
Change in exercise BP and maximum maximum exercise capacity | 6 months after randomization
  Change in exercise BP between baseline and 6 months and maximum exercise capacity between baseline and 6 months (difference between RDN and sham)
Change in Minnesota living with heart failure questionnaire (difference between RDN and sham) | 6 months after randomization
  Change in Minnesota living with heart failure questionnaire (difference between RDN and sham)
Change in Minnesota living with heart failure questionnaire | 6, 12 and 24 months after RDN
  Change in Minnesota living with heart failure questionnaire, compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Karl Fengler, PhD, Study Chair — Herzzentrum Leipzig, Universitätsklinik für Kardiologie
Locations (5):
- Germany (5):
  - Universitätsklinikum Halle (Saale), Klinik und Poliklinik für Innere Medizin III, Halle, Saxony-Anhalt
  - BG Klinikum Unfallkrankenhaus Berlin gGmbH, Berlin
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Kardiologie, Leipzig
  - Herzzentrum Leipzig, Universitätsklinik für Kardiologie, Leipzig
  - Universitätsmedizin der Johannes Gutenberg Universität Mainz, Zentrum für Kardiologie / Kardiologie 1, Mainz

IPD SHARING:
Plan to Share IPD: Yes
After publication of the major results and upon reasonable request from researchers performing an individual patient data meta-analysis, individual patient data that underlie published results will be shared after de-identification. This requires approval by the local Institutional Review Board (IRB) of the researcher requesting the data along with public registration of the meta-analysis.
  Summary statistics that go beyond the scope of published material will be made available to researchers for meta-analysis upon reasonable request and if the necessary data analysis is not unduly time-consuming. Together with publication of the main results, the trial protocol in full will be made publically available as well as the statistical analysis plan.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after publication of the major results